CLINICAL TRIAL: NCT01002027
Title: Models of Care: Evaluating a Best Practice Model of Treating Postnatal Depression (PND)
Brief Title: Three Model Care Pathways for Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Beyondblue (The National Depression Initiative) (Other)
Responsible Party: Jeannette Milgrom, University of Melbourne & Austin Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2005/01895
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Postnatal Depression
Keywords: Postnatal Depression; CBT-Counselling; Primary care
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT-counselling with Nurse (Active Comparator): CBT-counselling with Maternal Health Nurse, adjunctive to management by general medical practitioner
  Interventions: Behavioral: CBT-Counselling
- CBT-Counselling by Psychologist (Active Comparator): CBT-counselling with Psychologist, adjunctive to management by general medical practitioner
  Interventions: Behavioral: CBT-Counselling
- Routine management (No Intervention): Ongoing management by general medical practitioner

INTERVENTIONS:
Behavioral: CBT-Counselling — Intervention entailed six sessions of counselling-CBT delivered either by a trained Nurse, or by a Psychologist. Sessions focussed on: psycho-education about PND, main issues of concern, assessment of symptom severity, problem solving. Behavioural interventions (pleasant activities, anxiety management, relaxation, relationship communication) were used together with cognitive interventions (understanding links between thoughts and feelings, increasing positive thoughts, challenging negative self-talk and unhelpful beliefs).
  Arms: CBT-Counselling by Psychologist; CBT-counselling with Nurse

SUMMARY:
The study evaluates three best-practice care pathways for postnatal depression (PND) by comparing sole General Practitioner (GP) management to GP management in combination with CBT-based counselling from either a Psychologist or a Maternal and Child Health Nurse (MCHN).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women at 3-months postpartum

Exclusion Criteria:

* Psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Clinical Depression Score | 8 weeks post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Milgrom, PhD, Principal Investigator — University of Melbourne & Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Milgrom J, Holt CJ, Gemmill AW, Ericksen J, Leigh B, Buist A, Schembri C. Treating postnatal depressive symptoms in primary care: a randomised controlled trial of GP management, with and without adjunctive counselling. BMC Psychiatry. 2011 May 27;11:95. doi: 10.1186/1471-244X-11-95. PMID 21615968